CLINICAL TRIAL: NCT03024164
Title: Stroke Registration of Young Adults in China
Acronym: REACH
Status: Recruiting | Type: Observational
Sponsor: Yi Yang (Other)
Collaborators: Jiujiang No.1 People's Hospital (Other); Dezhou People's Hospital (Other); The Affiliated Hospital of Yanbian University (Other); First Affiliated Hospital of Jiamusi University (Unknown); Xuchang Central Hospital (Unknown); Inner Mongolia People's Hospital (Other); Shaoxing People's Hospital (Other); Chinese PLA General Hospital (Other); General Hospital of Ningxia Medical University (Other); General Hospital of Shenyang Military Region (Other); Siping Central People's Hospital (Other); The First Affilated Hospital of the Medical College, Shihezi University (Unknown); Daqing Oilfieled General Hospital (Unknown); Heilongjiang Provicial Hospital (Unknown); The First Affiliated Hospital of Soochow University (Other); Luoyang Central Hospital Affilated to Zhengzhou University (Unknown); Wuzhou Red Cross Hospital (Other); Cangzhou Central Hospital (Other); Binzhou Medical University (Other); Affilated Hospital of Inner Mongolia University for the Nationalities (Unknown); Fudan University Pudong Medical Center (Unknown)
Responsible Party: Sponsor-Investigator, Yi Yang, Associate dean, Director of Cerebrovascular Disease Center, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Other Study IDs: REACH
Record Dates: First submitted 2017-01-15; First posted 2017-01-18 (Estimated); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Ischemic Stroke
Keywords: youth; etiology; prognosis; recurrence; biomarkers
MeSH Terms: conditions — Ischemic Stroke; Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — EDTA-blood and serum will be collected for future analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Young adult stroke patients: Young adult (18-45 years old) patients with confirmed first-ever acute ischemic stroke
  Interventions: Other: Treatment following current guidelines

INTERVENTIONS:
Other: Treatment following current guidelines — Treatment following current guidelines

SUMMARY:
This is a multi-center, prospective,continuous registry study. The investigators will include 3000 young adult (18-45 years old) patients with confirmed first-ever acute ischemic stroke in China. The main purpose of this study is to build the study cohort of young ischemic stroke patients in China, and to compare the prognosis and stroke recurrence of young patients with different ischemic stroke subtypes. Secondary objectives are trying to find biomarkers of stroke recurrence.

DETAILED DESCRIPTION:
Approximately 10%-14% of all ischemic strokes occur in young adults ages 18 to 45 years old. Stroke etiology in this population differs by geographic region and has greater heterogeneity than in older individuals. Ascertain the definite etiologic classification in this young patients might be the key point to prevent the stroke recurrence and reduce the stroke burden. Advances in stroke diagnostic tests, particularly neuroimaging, refinement in classification schema. In this multi-center registry study conducted in China, we determine to explore the difference of prognosis and stroke recurrence of young patients with different ischemic stroke subtypes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 45 years, both genders
* First-ever acute ischemic stroke
* Onset of symptoms within 72 hours of inclusion
* Willing to participate in follow-up visits

Exclusion Criteria:

* Silent stroke
* Failure to give their informed consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young adult patients who had their first-ever ischemic stroke symptoms within 72 hours and visited one of the 22 participating medical centers in People's Republic of China.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-11-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Stroke recurrence | 1 year
  Percentage of patients with the 1 year new vascular events, defined as any event of the following: Any stroke (ischemic or hemorrhage)
Post-stroke disability | 3 months
  Modified Rankin Scale score changes (continuous) and dichotomized at percentage with score 0-2 vs. 3-6 at 3-month follow-up.

SECONDARY OUTCOMES:
Cardiovascular death | 3 months, 6 months and 1 year
  Percentage of patients with the 3-month, 6-month and 1 year cardiovascular death caused by any event of the following: Any stroke (ischemic or hemorrhage), sudden cardiac death, acute myocardial infarction, heart failure, and other cardiovascular death including pulmonary embolism, rupture of aortic aneurysm, cardiovascular interventional therapy, and peripheral arterial disease.
Other cardiovascular event | 3 months, 6 months and 1 year
  Percentage of patients with the 3-month, 6-month and 1 year other cardiovascular event including non-lethal myocardial infarction, and non fatal heart failure.
Other systemic embolism | 3 months, 6 months and 1 year
  Percentage of patients with the 3-month, 6-month and 1 year other systemic embolism except for cerebral artery, coronary artery, and pulmonary artery. Such as mesenteric arterial embolism,splenic artery embolization.

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No